CLINICAL TRIAL: NCT02921737
Title: A Phase II Trial of TAS-102 (Lonsurf) in Patients With Metastatic or Locally Advanced Unresectable Pancreatic Adenocarcinoma After Progression Through First Line Chemotherapy
Brief Title: TAS-102 (Lonsurf) in Metastatic or Locally Advanced Unresectable Pancreatic Adenocarcinoma Post First Line Chemotherapy (UF-STO-PANC-003)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient time to accrue sufficient subjects before end of funding
Sponsor: University of Florida (Other)
Collaborators: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601319 -A; UF-STO- PANC-003 (Other: University of Florida); IIT-USA-0115 (Other: Taiho Oncology); OCR15253 (Other: University of Florida)
Record Dates: First submitted 2016-09-26; First posted 2016-10-03 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Cancer
Keywords: metastatic; pancreatic; adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Adenocarcinoma | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): TAS-102
  Interventions: Drug: TAS-102

INTERVENTIONS:
Drug: TAS-102 — TAS-102 (35 mg/m2/dose) orally 2 times daily beginning the morning of Day 1 of each cycle and ending the evening of Day 5 of each cycle, as well as beginning the morning of Day 8 and ending the evening of Day 12 of each cycle. No TAS-102 will be given on Days 6-7 or Days 13-28 of each cycle.
  Other Names: Lonsurf

SUMMARY:
This is an open-label, non-randomized, sequentially enrolling single arm phase II trial to evaluate the activity of TAS-102 in previously treated metastatic and locally advanced unresectable pancreatic cancer after progression through or intolerance to first or second line chemotherapy. Trial therapy will consist of TAS-102 (Lonsurf®) 35 mg/m2 to be given orally twice daily on days 1-5 and 8-12 with cycles repeating every 28 days. The primary endpoint is to determine the progression free survival (PFS) in subjects with unresectable pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of adenocarcinoma of the pancreas, with pathologic confirmation of adenocarcinoma.
* Measurable disease per RECIST 1.1 criteria
* Metastatic or locally advanced unresectable disease. Subjects without clear evidence of distant metastatic disease will be presented at multidisciplinary tumor board for discussion of disease resectability.
* Refractory or intolerant to 1 or 2 prior regimens of standard chemotherapy for metastatic or locally advanced pancreatic cancer
* TAS102 will be planned to start after disease progression on first-or second line chemotherapy, provided any prior chemotherapy-related toxicities have resolved to less than or equal to Grade 1 or baseline within 28 days of the date the subject signs the informed consent form. Grade 2 or greater toxicities including alopecia, skin pigmentation,and platinum induced neurotoxicity/neuropathy are acceptable for starting on trial, as these toxicities do not preclude treatment with TAS102
* ECOG Performance Status of 0-2
* Capacity to understand and sign the informed consent document
* Able to take medications orally
* Life expectancy at least 12 weeks
* Age at least 18 years
* Patients on anticoagulation need to have no evidence of uncontrolled bleeding and be on a stable anticoagulation dose for at least 2 weeks prior to the date the subject starts study drug.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 3 months after the last dose of study drug to minimize the risk of pregnancy. Prior to signing the informed consent form, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
* WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as:

  * Amenorrhea that has lasted for ≥ 12 consecutive months without another cause, or
  * For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.

    * Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 3 months following the last dose of study drug.
    * Baseline laboratory values (bone marrow, renal, hepatic) must include:
* Adequate bone marrow function:

  1. Absolute neutrophil count >1500/mm3
  2. Platelet count >75,000/mm3
  3. HGB equal to or greater than 7g/dL
* Renal function:

  a. Serum creatinine ≤ 1.5 mg
* Hepatic function:

  1. Total bilirubin ≤ 1.5 mg/dL
  2. AST and ALT equal to or less than 3 times the upper limit of normal for patients without hepatic involvement, or AST and ALT equal to or less than 5 times the upper limit of normal for patients with hepatic involvement
  3. Serum calcium ≤ 12 mg/dl

Exclusion Criteria:

* Pregnant or lactating females
* Previously taken TAS-102
* Myocardial infarction or ischemia within the 6 months before first dose of study drug
* Uncontrolled' clinically significant dysrhythmia
* Intervention for ascites or pleural effusions within 4 weeks before first dose of study drug
* Previous surgery and/or radiotherapy may have been performed 2 or more weeks prior to the date the subject starts study treatment, provided that it was to a non-target lesion and there is still evidence of target lesion disease progression radiographically or intolerance to first- or second-line chemotherapy.
* Major surgery within 4 weeks before first dose of study drug (the surgical incision should be fully healed prior to study medication administration).
* Any anticancer therapy within 3 weeks before first dose of study drug.
* Extended field radiation within 4 weeks before first dose of study drug or limited field radiation within 2 weeks before first dose of study drug.
* Any investigational agent received within prior 4 weeks before first dose of study drug
* Subjects must not have more than one active malignancy at the time of enrollment
* Unresolved NCI-CTCAE toxicity grade 2 or higher attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation, and platinum induced neurotoxicity)
* Any co morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications including but not limited to chronic infections, uncontrolled diabetes, congestive heart failure according to the NYHA criteria, untreated brain metastases, liver or renal failure, gastrointestinal hemorrhage.
* Known untreated or unstable brain metastases or leptomeningeal disease
* Active infection
* Prisoners or subjects who are involuntarily incarcerated or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-07-26 (Actual); Study Completion 2020-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M. Duff, MD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - UF Health Cancer Center, Gainesville, Florida
  - Tallahasee Memorial HealthCare, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: To determine the progression free survival (PFS), which is defined as the duration of time from study entry to disease progression, death, or the date of last contact, whichever occurred first. Subjects were not included in the data for this outcome measure if they went off study for reasons other than disease progression, death or being lost to follow-up.
Time Frame: up to 54 weeks
Population: Only 6 subjects met the criteria to be included in the data for this endpoint.
Measure: Mean (Full Range); unit: weeks
Arm/Group | Treatment Arm
Number analyzed (Participants) | 6
weeks | 13.64 [0.14 to 53.86]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: To determine the objective response rate (ORR) by RECIST (Response Evaluation Criteria In Solid Tumors Criteria) v1.1 criteria. ORR is defined as the percentage of subjects who attained either a complete or partial response (CR + PR) by RECIST v1.1 criteria. RECIST v1.1 criteria defines a partial response (PR) as a decrease of the sum of the largest diameters of each target lesion by at least 30%. A complete response (CR) is defined as the disappearance of all target lesions (except lymph nodes, whose short axis must measure 10 mm or less).
Time Frame: 6 months
Population: Only two subjects were considered evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Clinical Benefit Rate
Description: To determine the Clinical Benefit Rate, defined as the percent of evaluable subjects who achieved either a complete or partial response or stable disease per RECIST v1.1 criteria. RECIST v1.1 criteria defines a partial response as a decrease of the sum of the largest diameter of each target lesion by at least 30%. A complete response is defined as the disappearance of all target lesions (except lymph nodes, whose short axis must measure 10 mm or less). By RECIST v1.1 criteria, a subject is considered to have stable disease when the sum of the largest diameter of the target lesions has neither decreased enough to qualify as a partial response not increased enough to qualify as progressive disease.
Time Frame: 6 months
Population: Only two subjects were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Time to Progression (TTP)
Description: To determine the time to progression (TTP), defined as the duration of time from study entry to disease progression
Time Frame: up to 54 weeks
Population: Disease progression only occurred for 5 subjects.
Measure: Mean (Full Range); unit: weeks
Arm/Group | Treatment Arm
Number analyzed (Participants) | 5
weeks | 15.43 [0.14 to 53.86]

5. Secondary Outcome: Overall Survival (OS)
Description: To determine overall survival (OS), defined as the duration of time from study entry to time of death.
Time Frame: up to 84 weeks
Measure: Mean (Full Range); unit: weeks
Arm/Group | Treatment Arm
Number analyzed (Participants) | 7
weeks | 23.45 [4.71 to 83.29]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at screening, on day 1 of each cycle, and up to 30 days after the last dose of study drug at a minimum, for up to 414 days.
Description: Adverse events were assessed by the principal investigator, the treating sub-investigator, and/or the study coordinator at screening, on day 1 of each treatment cycle, and up to 30 days after the last dose of study treatment at a minimum, for up to 414 days. Adverse events were assessed by physical examination, labs, and subject self-reports.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 7/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=7)
Hypokalemia (Metabolism and nutrition disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=7)
Abdominal pain (Gastrointestinal disorders) | 3
Alkaline phophatase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 5
Fever (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
diverticulitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neutrophil count decreased (Investigations) | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
White blood cell count decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT02921737/Prot_SAP_000.pdf